CLINICAL TRIAL: NCT03668938
Title: Efficacy of Occupational Therapy in the Rehabilitation of Complex Patients: Randomized Controlled Trial
Brief Title: Occupational Therapy Intervention in Patients With Complex Needs to Improve Social Reintegration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COMPLE-TO_2018
Record Dates: First submitted 2018-08-14; First posted 2018-09-13 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2022-07

CONDITIONS: Rehabilitation; Occupational Therapy
Keywords: Occupational Therapy; Complex Patient; Randomized Control Trial; Social Reintegration
MeSH Terms: interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: masking of outcome assessor to T0
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental): The occupational therapy intervention provides a treatment aimed at improving autonomy in the activities chosen by the patient
  Interventions: Other: Occupational Therapy; Other: usual care
- usual care (Active Comparator): Usual care consists in rehabilitation treatment delivered by a multidisciplinary team
  Interventions: Other: usual care

INTERVENTIONS:
Other: Occupational Therapy — The intervention in the hospitalization phase is mainly aimed at achieving the objectives related to the self-care area and, secondly, to the objectives in the areas of productivity and leisure time, identified in T0 and to the environmental assessment of the places of life of the patient; more an intervention in the patient's post-discharge home, mainly aimed at achieving the objectives related to social reintegration, the area of productivity and leisure time and, secondly, to possible objectives in the areas of self-care identified in T1.
  Arms: intervention
Other: usual care — Usual care consists in rehabilitation treatment delivered by a multidisciplinary team

SUMMARY:
A previous study that involved the intervention of the occupational therapist (OT) on complex patients both in hospital and at home showed the effectiveness of OT during hospitalization. The effectiveness was not demonstrated in the post-discharge phase. Now, the investigators presented a RCT to compare the levels of social reintegration between the intervention group and control group. The hypothesis is that the intervention group obtains a higher and clinically relevant level of social reintegration compared to the group treated with the usual care.

DETAILED DESCRIPTION:
In the previous study, the intervention group achieved higher gains in the return to normal life than in the control group, but this difference did not reach statistical significance. Because of this, a new study was implemented with the correct sample size, defined through the previous study. In addition, the post-discharge phase the COPM was administered to define new objectives relating mainly to productivity and leisure time areas. Finally, the investigators have indentified some territorial services with the aim to create tailored paths/interventions for patients to promote social reintegration.

ELIGIBILITY:
Inclusion Criteria:

* Complex impatient
* Admitted to AUSL-IRCCS/UO MFR

Exclusion Criteria:

* Language barriers
* Severe cognitive impairment
* Psychiatric disorders
* Domiciled in a protected facility at the time of admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Change in Reintegration to Normal Living Index | Time 1 is on average 45 days from Time 0 (discharge from the rehabilitation ward); Time 2 is at 90 days ± 15 days from discharge
  Compare the change in the level of reintegration to normal life between the two arms. The score range is from 1 to 100. Higher values represent a better outcome.

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure | Time 0 is the baseline at the patient ammission in the rehabilitation ward; Time 1 is on average 45 days from Time 0 (discharge from the rehabilitation ward); Time 2 is at 90 days ± 15 days from discharge
  Compare the results obtained in the two groups in the performance and satisfaction perceived by the patient in carrying out the occupational activities identified as priorities. The score range is from 1 to 10. Higher values represent a better outcome.
Modified Barthel Index | Time 0 is the baseline at the patient ammission in the rehabilitation ward; Time 1 is on average 45 days from Time 0 (discharge from the rehabilitation ward); Time 2 is at 90 days ± 15 days from discharge
  Compare the results obtained in the two groups in autonomy in the activities of daily life. The score range is from 1 to 100. Higher values represent a better outcome.
Instrumental Activity of Daily Living | Time 0 is the baseline at the patient ammission in the rehabilitation ward; Time 1 is on average 45 days from Time 0 (discharge from the rehabilitation ward); Time 2 is at 90 days ± 15 days from discharge
  Compare the results obtained in the two groups in autonomy in instrumental activities. The score range is from 1 to 8. Lower values represent a better outcome.
Hospital Anxiety and Depression Scale | Time 0 is the baseline at the patient ammission in the rehabilitation ward; Time 1 is on average 45 days from Time 0 (discharge from the rehabilitation ward); Time 2 is at 90 days ± 15 days from discharge
  Compare the results obtained in the two groups in anxiety and depression.The scale has 2 subscales that evaluates anxiety and depression, respectively. For both subscales the score range is from 0 to 21. Higher values represent a better outcome.
Short Form 12 | Time 1 is on average 45 days from Time 0 (discharge from the rehabilitation ward); Time 2 is at 90 days ± 15 days from discharge
  Compare the results obtained in the two groups in the quality of life. The scale has 2 subscales. The Physical Component Summary has a score range from 11 to 70. The other subscale evaluates the Mental Component Summary with a score range from 7 to 72. Higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Fugazzaro, Principal Investigator — Local Health Autority of Reggio Emilia
Locations (1):
- Ospedale Santa Maria Nuova, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costi S, Pellegrini M, Braglia L, Cavuto S, Fugazzaro S. Occupational therapy improves social participation of complex patients discharged from hospital: results of a powered randomized controlled trial. Disabil Rehabil. 2024 Jun;46(11):2223-2233. doi: 10.1080/09638288.2023.2218653. Epub 2023 Jun 1. PMID 37259592